CLINICAL TRIAL: NCT07019363
Title: A Study on the Efficacy and Safety of CDK4/6 Inhibitors Combined With Standard Adjuvant Endocrine Therapy in High-Risk, HR+/HER2+ Early Breast Cancer Patients Who Have Completed Adjuvant Anti-HER2 Targeted Therapy"
Brief Title: CDK4/6 Inhibitors Combined With Standard Adjuvant Endocrine Therapy in High-Risk, HR+/HER2+ Early Breast Cancer Patients(CHESS)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Director of General Surgery of Fudan Shanghai Cancer Center, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCHBCC-N091
Record Dates: First submitted 2025-05-04; First posted 2025-06-13 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer; Adjuvant Therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen; Anastrozole; Letrozole; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): endocrine therapy
  Interventions: Drug: Endocrine Therapy (Tamoxifen, Anastrozol, Letrozole, Exemestane)
- Experimental (Experimental): Standard endocrine therapy combined with CDK4/6i
  Interventions: Drug: Standard endocrine therapy combined with CDK4/6 Inhibitor

INTERVENTIONS:
Drug: Endocrine Therapy (Tamoxifen, Anastrozol, Letrozole, Exemestane) — Standard endocrine therapy
  Arms: Control
Drug: Standard endocrine therapy combined with CDK4/6 Inhibitor — CDK4/6 inhibitor therapy for 2 years in combination with standard endocrine therapy
  Arms: Experimental

SUMMARY:
This study is a prospective, open-label, multicenter, randomized controlled Phase III clinical trial. Building upon anti-HER2 targeted therapy combined with endocrine therapy, the addition of CDK4/6 inhibitors has demonstrated greater clinical benefits for advanced TPBC patients. This study aims to investigate the efficacy and safety of CDK4/6 inhibitor combination with standard adjuvant endocrine therapy in HR+/HER2+ early breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Females aged ≥18 and ≤70 years.
2. ECOG systemic status grade 0 to 1.
3. Histologically confirmed invasive HR+/HER2+ breast cancer (Specific definition: breast cancer patients whose estrogen receptor (ER), progesterone receptor (PR), and human epidermal growth factor receptor 2 (HER-2) are all determined to be positive by pathologic testing. Specifically: ER positive: IHC>10%, PR positive: IHC>10%, HER2 positive: IHC+++ or IHC++ but amplified by FISH.
4. Early-stage breast cancer after radical mastectomy with postoperative pathology consistent with TNM staging of ≥pN1 ; or postoperative pathology suggestive of non-pCR after neoadjuvant therapy; or postoperative pathology suggestive of pCR after neoadjuvant therapy but with clinical staging consistent with cT4 or N3 before neoadjuvant therapy
5. Within 1 year of completion of adjuvant anti-HER2 targeted therapy: anti-HER2 targeted therapy includes trastuzumab-based therapy, and/or T-DM1 therapy, and/or TKI therapy.
6. The function of major organs is basically normal, and the following conditions are met: ① The criteria for routine blood tests need to be met: HB ≥ 90g/L (no blood transfusion within 14 days); ANC ≥ 1.5 × 109/L; PLT ≥ 75 × 109/L; ② The biochemical tests need to be met as follows: TBIL ≤ 1.5 × ULN (the upper limit of normal value); ALT and AST ≤ 3 × ULN; serum Cr ≤ 1 × ULN, and endogenous creatinine clearance > 50 ml/min (Cockcroft-Gault formula).
7. Female subjects of childbearing potential are required to use a medically approved form of contraception during study treatment, and for at least 3 months after the last dose of study drug.
8. Subjects voluntarily enrolled in the study, signed an informed consent form, were compliant, and cooperated with follow-up visits.

Exclusion Criteria:

1. Bilateral breast cancer;
2. Metastasis to any site;
3. Taking food or medications that are strong inhibitors or inducers of CYP3/4.

   1. Strong inhibitors of CYP3/4 include: boceprevir, clarithromycin, konifactam, delavirdine, indinavir, itraconazole, ketoconazole, ritonavir, mibefradil, miconazole, fazodone, nelfinavir, propoxiconazole, ritonavir, saquinavir, naloxone, telaprevir, telithromycin, voriconazole, grapefruit, grapefruit juice, or grapefruit containing foods.
   2. Strong inducers of CYP3/4 including carbamazepine, phenytoin, pramipexole, rifampin, and St. John's wort.
4. History of clinically significant or uncontrolled cardiac disease including congestive heart failure, angina pectoris, myocardial infarction within the last 6 months, or ventricular arrhythmia;
5. other malignancy within the previous 5 years, excluding cured carcinoma in situ of the cervix, basal cell carcinoma of the skin, or squamous cell carcinoma of the skin;
6. Pregnant or lactating women, women of childbearing age who are unable to use effective contraception;
7. Patients who are concurrently enrolled in other clinical trials;
8. severe or uncontrolled infection;
9. Patients with known active HBV or HCV infection or Hepatitis B DNA ≥500, or chronic stage with abnormal liver function;
10. Those with a history of psychotropic substance abuse that cannot be stopped or those with psychiatric disorders;
11. Patients who, in the judgment of the investigator, are not suitable for participation in this study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1903 (Estimated)
Dates: Start 2025-06-15 (Actual); Primary Completion 2029-05-15 (Estimated); Study Completion 2033-04-15 (Estimated)

PRIMARY OUTCOMES:
5-years Invasive disease free survival | 5 years
  5-year invasive disease-free survival (iDFS), defined as the time from randomization to the first occurrence of: local recurrence, distant metastasis, contralateral invasive breast cancer, death from any cause.

SECONDARY OUTCOMES:
Distant Recurrence-Free Survival (DRFS) | 5 years
  DRFS is defined as the time interval from the start of cancer treatment to the first occurrence of distant metastasis or death from any cause.
Overall Survival (OS) | Approximately 5 years
  OS is defined as the time from randomisation until the date of death due to any cause.
Safety including adverse events (AEs), severe adverse events (SAEs) and adverse events of special interest (AESI). | Up to approximately 3 years
  Incidence of AEs, SAE, AESIs (interstitial lung disease, LVEF decrease), AEs resulting in study intervention interruption and discontinuation, etc.
Patient-Reported Outcome (PRO) | Up to approximately 3 years
  Patient-Reported Outcome (PRO) refers to a report that comes directly from the patient on her health status, functional status, and experience of treatment, without interpretation by healthcare or other personnel (e.g., symptoms, quality of life, physical functioning, etc.), and is usually collected through standardized questionnaires or scales. Lower scores in European Organization for Research and Treatment of Cancer(EORTC) QLQ-BR45 questionnaire will mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: zhimin shao, Principal Investigator — Fudan University
Locations (1):
- Fudan cancer center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No